CLINICAL TRIAL: NCT01771523
Title: Is the Use of Drain for Thyroid Surgery Realistic?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, manuk norayk manukyan, Associated Professor, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: mütf2
Record Dates: First submitted 2011-08-03; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Goiter
Keywords: thyroidectomy; drain use
MeSH Terms: conditions — Goiter | interventions — Thyroidectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): thyroidectomy
  Interventions: Procedure: Thyroidectomy
- Group 2 (Active Comparator): thyroidectomy use of drain
  Interventions: Procedure: Thyroidectomy; Device: use of drain

INTERVENTIONS:
Procedure: Thyroidectomy — total thyroidectomy or lobectomy
Device: use of drain — drain will be used
  Arms: Group 2

SUMMARY:
Background : The use of suction drains in thyroid surgery is common practice in order to avoid haematoma or seroma, as well as to identify promptly the onset of haemorrhaging that might compromise the patient's airway. The aim of this study to determine the effects of routine drainage compared to no drainage in thyroidectomy patients.

Study Design : Total of 400 patients who undergoing total thyroidectomy or lobectomy for thyroidal disorders will be randomly allocated to be drained or not. Postoperative ultrasonographic (USG) neck examination will be performed for all patients on postoperative 24th hour by the same ultrasonologist each time. Postoperative pain, complications and hospital stay will be recorded. The statistical analysis will be performed and p<0,05 will be accepted as an important statistical value (SPSS 16.0 for Windows).

DETAILED DESCRIPTION:
Patients will include in the study will randomly allocate to drain and non-drain group on the basis of computer generated random number table. Patients with substernal goitre or non differentiated cancer will exclude from the study.

According to the thyroidal disorder, total thyroidectomy or lobectomy plus isthmectomy will be performed. The operating time will be defined as the time from the first incision to the last suture's placement. 4/0 polypropylene sutures will be used subcutaneously for wound closure. In the drain group a closed suction drain with negative pressure (Hemovac®) was brought out through a separate wound.

ELIGIBILITY:
Inclusion Criteria:

* All patients required thyroidectomy

Exclusion Criteria:

* Patients with substernal goitre or non differentiated cancer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Postoperative fluid accumulation (ml.) | Postoperative first 24 hours
  Standard thyroidectomy is proven method for safety. We will perform standard thyroidectomy in this study. In this period, patients will be monitored for bleeding and seroma. Major bleeding rare complication for thyroid surgery but requires re-operation immediately. Many studies suggested that drains may block with clotted blood and do not alert the surgeon, even if major bleeding occurs(1,2,3). We don't use drain routinely in standard thyroidectomy in our clinic for seven years. Bleeding and reoperation rates are similar between the literature and our clinic. The amount of fluid collection in thyroid bed will be assessed by Ultrasonography in postoperative 24th hours. Volume of fluid collection in the operative bed will be calculated by measuring the maximum diameter in three dimensions.Similar results between groups are evidence that the use of drain is not necessary.

SECONDARY OUTCOMES:
Postoperative pain score on the visual analog scale (0-10) | 6th hours and 24th hours
  Postoperative pain will be assessed according to a visual analogue scale (VAS) from 0 (no pain) to 10 (worst pain imaginable) on the postoperative sixth hour (POSH-VAS) and postoperative first day (POFD-VAS).The mean VAS scores will be compared drain and non-drain group.

OTHER OUTCOMES:
Number of postoperative complications. | postoperative first 6th hour, 24th hour, third day, third month, sixth month, first year
  We will demonstrate there was no significant differences in postoperative complications between subgroups.Similar complications rates will be demonstrate absence of drains for thyroid surgery is safe and efficient.
Length of hospital stay | postoperative period (days)
  Use of drain increases length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Deveci, Ass. Prof., Principal Investigator — Maltepe University, School of Medicine , General Surgery Department; Manuk N. Manukyan, Ass.Prof., Study Director — Maltepe University, School of Medicine, General Surgery Department; Abut Kebudi, Prof., Study Chair — Maltepe University, School of Medicine, General Surgery Department; Fatih Altintoprak, Ass.Prof., Principal Investigator — Sakarya University, School of Medicine, General Surgery Department; Neşe Yener, Ass.Prof., Principal Investigator — Maltepe University, School of Medicine, Pathology Department; Sertan Kapakli, Ass.Prof., Principal Investigator — Maltepe University, School of Medicine, General Surgery Department; Rahmi Çubuk, Ass.Prof., Principal Investigator — Maltepe University, School of Medicine, Radiology Department
Locations (1):
- Maltepe University School of Medicine, General Surgery Department, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Deveci U, Altintoprak F, Sertan Kapakli M, Manukyan MN, Cubuk R, Yener N, Kebudi A. Is the use of a drain for thyroid surgery realistic? A prospective randomized interventional study. J Thyroid Res. 2013;2013:285768. doi: 10.1155/2013/285768. Epub 2013 May 30. PMID 23819100
- See also: Thyroid surgery without drainage: 15 years of clinical experience. — http://www.ncbi.nlm.nih.gov/pubmed?term=Arriyanayagam%20DC%2C%20Narayan%20Singh%20V%2C%20Busby%20D%2C%20Sieunarine%20K%2C%20Raju%20G%3A%20Thyroid%20surgery%20without%20drainage%3B%2015%20years%20of%20clinical%20experience.%20Journal%20of%20Royal%20
- See also: Is the routine drainage after surgery for thyroid necessary? A prospective randomized clinical study [ISRCTN63623153]. — http://www.ncbi.nlm.nih.gov/pubmed/15946379
- See also: Drainage after total thyroidectomy or lobectomy for benign thyroidal disorders. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2276675/